CLINICAL TRIAL: NCT07396038
Title: Evaluation of Intraoperative Bladder Injuries During Transurethral Resection of Bladder Tumors Using the BICEP Classification (BICEP on TURBT)
Brief Title: INTRAOPERATIVE BLADDER INJURY ASSESSMENT IN TURBT USING BICEP
Acronym: BICEP in TURBT
Status: Not yet recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); Medical University of Graz (Other); Hannover Medical School (Other); King's College London (Other)
Responsible Party: Principal Investigator, Selim Soyturk, Urologist / Coordinating Investigator, Necmettin Erbakan University
Other Study IDs: ReScore26-1
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer; TURBT; Bladder Injury
Keywords: Transurethral resection of bladder tumor; Bladder perforation; Bladder cancer surgery; Bladder injury classification; Ureteral orifice injury; Endoscopic bladder surgery complications
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TURBT PATIENT COHORT: Patients undergoing transurethral resection of bladder tumor for diagnostic, staging, primary treatment, or re-resection purposes. All participants are evaluated intraoperatively for the presence and severity of bladder injuries using a standardized endoscopic injury classification system, with subsequent recording of perioperative and early postoperative outcomes.
  Interventions: Other: No intervention is assigned as part of this observational study. All procedures are performed as part of routine clinical care.

INTERVENTIONS:
Other: No intervention is assigned as part of this observational study. All procedures are performed as part of routine clinical care. — No intervention is assigned as part of this observational study. All procedures are performed as part of routine clinical care.

SUMMARY:
Transurethral resection of bladder tumor (TURBT) is the cornerstone procedure in the diagnosis and treatment of bladder cancer but is associated with a spectrum of intraoperative bladder injuries ranging from minor mucosal tears to major perforations. Currently, there is no standardized intraoperative classification system specifically designed to grade and report these injuries during TURBT.

This study aims to apply the Bladder Injury Classification System for Endoscopic Procedures (BICEP) to TURBT in order to systematically classify intraoperative bladder injuries, evaluate their management, and explore their association with perioperative and early postoperative outcomes.

DETAILED DESCRIPTION:
Transurethral resection of bladder tumors (TURBT) is a fundamental endourological procedure for the diagnosis, staging, and initial management of bladder cancer. Despite its widespread use and standardized oncological objectives, TURBT is associated with a broad spectrum of intraoperative bladder injuries, ranging from minor mucosal lesions to major bladder perforations or ureteral orifice injuries. Currently, intraoperative bladder injuries during TURBT are inconsistently defined and reported, often being retrospectively captured only through postoperative complication grading systems, which limits objective comparison between techniques, surgeons, and centers.

This study is designed as an observational patient registry aiming to systematically evaluate intraoperative bladder injuries occurring during TURBT using the Bladder Injury Classification System for Endoscopic Procedures (BICEP). The BICEP classification is an anatomically based intraoperative grading system that categorizes bladder injuries according to depth, severity, and required management, allowing standardized real-time documentation of endoscopic injuries. By applying this framework to TURBT, the registry seeks to establish a reproducible and clinically meaningful method for injury reporting in oncologic endourology.

The registry will prospectively collect perioperative data from patients undergoing TURBT, including tumor characteristics, operative setting, energy modality, resection technique, intraoperative events such as obturator reflex, and bleeding severity. Intraoperative bladder injuries will be classified using the predefined BICEP categories, and injury timing, anatomical location, confirmation methods, and management strategies will be recorded in a structured manner. Postoperative clinical course data will be captured to allow assessment of early outcomes and short-term clinical impact.

This registry is implemented using a standardized electronic data capture system with predefined variable definitions and structured fields. Data quality is ensured through built-in range checks, mandatory fields for key variables, and internal consistency rules to minimize incomplete or conflicting entries. A detailed data dictionary defines each variable, its clinical meaning, coding structure, and acceptable value ranges to ensure uniform interpretation across participating centers. Source data for registry entries are derived from routine clinical documentation, including operative reports, anesthesia records, and postoperative follow-up notes.

Participating centers are instructed to enter consecutive eligible cases to reduce selection bias and improve representativeness. Periodic data reviews are planned to assess completeness, logical consistency, and adherence to registry definitions. Data validation procedures include cross-checks between related variables (for example, injury grade and management strategy) to identify discrepancies. The registry is designed to be expandable, allowing future linkage with additional outcomes or long-term oncological follow-up modules if required.

Sample size is not fixed a priori, as the registry is designed to capture real-world practice patterns and complication profiles across centers. Accrual will continue until a sufficient number of cases is obtained to allow meaningful descriptive and comparative analyses of injury patterns and associated perioperative factors. Missing data will be handled using predefined categories (unknown, not applicable) and will be reported transparently in analyses.

Statistical analysis will primarily focus on descriptive statistics to characterize injury incidence and severity, followed by exploratory analyses evaluating associations between intraoperative bladder injury grades and perioperative variables or early postoperative outcomes. Analytical methods will be aligned with the observational nature of the registry and hypothesis-generating intent of the study.

By establishing a structured and standardized registry for intraoperative bladder injuries during TURBT, this study aims to improve the quality of complication reporting, facilitate comparison between surgical techniques and energy modalities, and provide a foundation for future prospective validation studies and quality improvement initiatives in endourological oncology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Patients undergoing transurethral resection of bladder tumor
* Procedures performed for primary resection, re-resection, diagnostic, or staging purposes

Exclusion Criteria:

* Patients with incomplete intraoperative data regarding bladder injury assessment
* Patients who decline participation, if informed consent is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing transurethral resection of bladder tumors at participating centers. Participants are identified from consecutive cases in which intraoperative bladder injury assessment is performed and recorded using a standardized classification approach during the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative bladder injury severity assessed using the BICEP classification | During the surgical procedure (intraoperative)
  Intraoperative bladder injuries occurring during transurethral resection of bladder tumors are classified and graded using the Bladder Injury Classification System for Endoscopic Procedures (BICEP), an ordinal scale ranging from 0 (no injury) to 4 (most severe injury requiring surgical intervention). Higher scores indicate greater injury severity.

SECONDARY OUTCOMES:
Characteristics of intraoperative bladder injuries | Intraoperative and immediate postoperative period
  Anatomical location, timing, and severity distribution of intraoperative bladder injuries as classified by the BICEP system.
Management of intraoperative bladder injuries according to BICEP grade | Intraoperative and immediate postoperative period
  Management strategies applied for intraoperative bladder injuries based on BICEP classification, including conservative management, prolonged catheterization, endoscopic intervention, or surgical repair.
Postoperative catheter duration | From end of surgery until catheter removal, up to 30 days postoperatively
  Duration of urinary catheterization following transurethral resection of bladder tumors in relation to BICEP classified intraoperative bladder injuries.
Length of hospital stay | From end of surgery until hospital discharge during index hospitalization (up to 30 days)
  Length of hospitalization following transurethral resection of bladder tumors according to the presence and severity of BICEP classified intraoperative bladder injuries.
Readmission within 30 days | 30 days postoperative
  Unplanned hospital readmission for any cause within 30 days after transurethral resection of bladder tumors in patients with and without BICEP-classified intraoperative bladder injuries.
Re-intervention within 30 days | 30 days postoperative
  Additional endoscopic or surgical interventions required within 30 days following transurethral resection of bladder tumors in relation to BICEP classified intraoperative bladder injuries.
Postoperative complications | 30 days postoperative
  Postoperative complications graded according to the Clavien Dindo classification system and analyzed in relation to BICEP classified intraoperative bladder injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Selçuk Güven, Prof, Study Chair — Necmettin Erbakan University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available upon reasonable request for research purposes. Data will be shared following local ethics committee approval and execution of a data-use agreement. No direct patient identifiers will be shared. Data will include demographic variables, baseline assessments, operative details, postoperative outcomes, and follow-up measures collected in the registry.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) and supporting documents will be available beginning 12 months after publication of the primary results manuscript and will remain available for a minimum of 5 years thereafter.
Access Criteria: only qualified researchers with a methodologically sound proposal will be granted access. Requests must be reviewed and approved by the principal investigator and require completion of a data-use agreement. Access will be provided in de-identified format only and delivered via secure, password-protected electronic transfer. No direct identifiers or protected health information will be shared.

REFERENCES:
- [Background] Breda A, Gallioli A, Diana P, Fontana M, Territo A, Gaya JM, Rodriguez-Faba O, Huguet J, Piana A, Verri P, Baboudjian M, Aumatell J, Algaba F, Palou J. The DEpth of Endoscopic Perforation scale to assess intraoperative perforations during transurethral resection of bladder tumor: subgroup analysis of a randomized controlled trial. World J Urol. 2023 Oct;41(10):2583-2589. doi: 10.1007/s00345-022-04052-w. Epub 2022 Jun 4. PMID 35665840
- [Background] Akgul B, Tozsin A, Tokas T, Micali S, Herrmann T, Bianchi G, Fiori C, Altinkaya N, Ortner G, Knoll T, Lehrich K, Bohme A, Gadzhiev N, Omar M, Kartalas Goumas I, Romero Otero J, Aydin A, Lusuardi L, Netsch C, Khan A, Greco F, Dasgupta P, Tunc L, Rassweiler J, Serdar Gozen A, Ahmed K, Guven S. Development of a Bladder Injury Classification System for Endoscopic Procedures: A Mixed-methods Study Involving Expert Consensus and Validation. Eur Urol Focus. 2025 Jan;11(1):126-135. doi: 10.1016/j.euf.2024.09.004. Epub 2024 Sep 25. PMID 39327217